CLINICAL TRIAL: NCT05507047
Title: The Evaluation of Enamel Matrix Derivative on the Bone Regenerative Potential of the Dental Implant With Transcrestal Sinus Lifting Technique: Randomized-Controlled CBCT Study
Brief Title: Emdogain Implementation With Transcrestal Sinus Lifting and Dental Implant Placement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: T.C. Dumlupınar Üniversitesi (Other)
Responsible Party: Principal Investigator, Berceste Guler, Assoc Prof, T.C. Dumlupınar Üniversitesi
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 14/4
Record Dates: First submitted 2022-08-15; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Osseointegration Failure of Dental Implant; Bone Density Increased
Keywords: enamel matrix derivated; maxillary sinus
MeSH Terms: conditions — Osteosclerosis | interventions — enamel matrix proteins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Transcrestal Sinus Lifting with Emdogain (Experimental): Osteotome sinus floor elevation with enamel matrix derivated
  Interventions: Drug: Enamel Matrix Protein
- Transcrestal Sinus Lifting (Active Comparator): Osteotome sinus floor elevation
  Interventions: Drug: Enamel Matrix Protein

INTERVENTIONS:
Drug: Enamel Matrix Protein — Enamel matrix derivated is used with transcrestal sinus lifting treatment
  Other Names: emdogain

SUMMARY:
The aim of this study is to evaluate the clinical and radiographic results of implants placed using osteotome sinus ﬂoor elevation (OSFE) with and without simultaneous enamel matrix derivative (EMD) application.

DETAILED DESCRIPTION:
Twenty-four patients will be randomly assigned into two groups: Group I: (EMD+OSFE) (n=20 implants, 13 patients) OSFE with EMD application, and Group II 8OSFE): (n=20 implants, 11 patients) OSFE without EMD application. The patients will be recall at 3- and 12- months after surgery. The residual bone height (RBH), implant protrusion length (IPL), peri-implant sinus bone level (SBL), endo-sinus bone gain (ESBG), implant stability and peri-implant bone density values (Hounsfield units) will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* partial edentulism in the maxillary posterior region for at least 4 months from tooth loss and require implant treatment
* adequate bone thickness for primary stabilization
* residual bone height ranged from 4 mm to 6 mm
* systemic and local conditions compatible with implant placement and sinus ﬂoor elevation
* antagonist teeth

Exclusion Criteria:

* uncontrolled diabetes mellitus or other systemic disorders (such as; hepatitis, tuberculosis, AIDS)
* pregnancy
* untreated periodontal disease
* endodontic lesions or other oral disorders
* heavy smokers (≥10 cigarettes per day)
* acute or chronic rhinitis
* sinusitis or pathology in sinus
* inadequate residual bone height and quality to achieve implant stability
* previous implant treatment/failure or bone augmentation in the implant site
* sinus perforation as confirmed via Valsalva maneuver
* insufficient primary implant stability measured by RFA

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-01 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
endo-sinus bone gain | CBCT will be evaluated at initiation of study (T0), at 3th month (T1) and 12th month (T2)
  New bone formation into sinus (NB) following OSFE- measured by endo-sinus bone gain

SECONDARY OUTCOMES:
radiographic measurements | CBCT will be evaluated at initiation of study (T0), at 3th month (T1) and 12th month (T2)
  The residual bone height (RBH)
implant stability | It will be measured at initiated at implant placement and third month follow-up
  resonance frequency analysis
Radiographic measurements | CBCT will be evaluated at initiation of study (T0), and at 12th month (T2)
  implant protrusion length into the sinus
peri-implant sinus bone level | CBCT will be evaluated at initiation of study (T0), at 3th month (T1) and 12th month (T2)
  the distance between the groove most coronal to the implant and the bone-implant connection most apical to the implant
Densitometric Analysis | Bone Density was measured at baseline, 3- and 12-months by CBCT scans
  CBCT allows sectional analysis. Each axial image is 260000 megapixels, and each pixel has a CT number (Hounsfield unit). The higher the CT number, the denser the object

CONTACTS AND LOCATIONS:
Overall Officials: Deniz Ozbay, DDS PhD, Principal Investigator — Gazi University
Locations (1):
- Gazi University Faculty of Dentistry, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Vincent-Bugnas S, Charbit Y, Charbit M, Dard M, Pippenger B. Maxillary Sinus Floor Elevation Surgery With BioOss Mixed With Enamel Matrix Derivative: A Human Randomized Controlled Clinical and Histologic Study. J Oral Implantol. 2020 Oct 1;46(5):507-513. doi: 10.1563/aaid-joi-D-19-00119. PMID 32299097
- See also: Maxillary Sinus Floor Elevation Surgery With BioOss Mixed With Enamel Matrix Derivative — https://pubmed.ncbi.nlm.nih.gov/32299097/
- See also: Effect of enamel matrix derivative on alveolar ridge preservation in the posterior maxilla — https://pubmed.ncbi.nlm.nih.gov/32902075/